CLINICAL TRIAL: NCT06017310
Title: Evaluation of the Type 1 IFN Response in Viral Infections
Brief Title: Respiferon Project
Acronym: Respiferon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0697
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Viral Infection
Keywords: respiratory viruses; Nasal IFN-1 Score; Nasopharyngeal Swab; Replicative virus; Infectiousness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Replicative viruses: Presence of a replicative virus determined by viral culture
  Interventions: Diagnostic Test: Evaluate the performance of IFN I/III
- Unreplicative viruses: Absence of a replicative virus determined by viral culture
  Interventions: Diagnostic Test: Evaluate the performance of IFN I/III

INTERVENTIONS:
Diagnostic Test: Evaluate the performance of IFN I/III — Evaluate the response in diagnosing non-respiratory viral infection.

SUMMARY:
Respiratory viral infections (RVIs) represent a major public health problem and a great burden in terms of morbidity and mortality in children and adults worldwide. To ascertain the source of an infection, microbiology laboratories routinely perform a crucial step: the search for the pathogen through Polymerase Chain Reaction (PCR). Due to the extensive variety of pathogens, testing for the existence of all potential viruses, bacteria, or fungi accountable for the infection is an impractical and time-intensive endeavor. Furthermore, the rise of novel pathogens, exemplified by those accountable for the recent SARS-CoV-2 pandemic, underscores the urgency of promptly developing new innovative diagnostic tests.

To address these needs, researchers have dedicated several years to developing indirect methodologies notably centered around utilizing markers derived from the host's immune system. Among these, one particularly promising approach focuses on measuring the expression of interferon-stimulated genes, which are uniquely triggered by viral infections, thereby facilitating viral diagnosis. This methodology's efficacy has been proven in the context of SARS-CoV-2 infections.

This study's objective is to assess the functionality of such a tool across a spectrum of Respiratory Viral Infections (RVIs) prevalent within a French population during the winter season.

ELIGIBILITY:
Inclusion Criteria:

* Positive nasopharyngeal samples for the detection of a virus, for which the replicative character has been established by the viral culture technique (500µL minimum required)
* Samples kept at the CRB since 2018
* Information to patients carried out and non-objection collected-

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized at the Hospices Civils de Lyon (HCL) with respiratory infection symptoms.
  Nasopharyngeal samples positive for the detection of a respiratory virus for which the viral culture has been carried out will be selected by the CRB. After informing the patients of the study, the IFN I/III response can be assessed on these same nasopharyngeal samples (no additional sample necessary).
  The data thus obtained will allow to determine the capacity of the IFN I/III response to detect replicating viruses.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence or Absence of a replicative virus detected by viral culture | One sample at inclusion
  RT-qPCR/qPCR-positive NPS will be inoculated on suitable cell lines using a culture medium appropriate for growth. Plates will be incubated at 33°C in 5% CO2 for 96 hours. Positive samples will be harvested for the confirmation technique, while negative samples will be cultured for 8 days. RNA or DNA from infected cells will be harvested and will be assayed with Panther Fusion® RT-PCR/PCR kits (Hologic Inc., San Diego, CA, USA) for viral identification, except for RSV and influenza A and B viruses (IAV/IBV) which were detected by immunofluorescence using Thermo ScientificTM IMAGENTM kits (Thermo Fischer Scientific, Waltham, MA, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Infective Agents Institute, Croix rousse Hospital, Lyon, Rhone, France